CLINICAL TRIAL: NCT03436563
Title: A Phase Ib/II Trial of M7824 in Solid Tumors With Microsatellite Instability With Consensus Molecular Subtype 4 Metastatic Colorectal Cancer in Combination With Radiation, or in Colorectal Cancer Patients With Detectable Circulating Tumor DNA Following Definitive Therapy
Brief Title: M7824 in Patients With Metastatic Colorectal Cancer or With Advanced Solid Tumors With Microsatellite Instability
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0339; NCI-2018-00919 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0339 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Colon Adenocarcinoma; High-Frequency Microsatellite Instability; Metastatic Malignant Solid Neoplasm; Rectal Adenocarcinoma; Refractory Colorectal Carcinoma; Stage IV Colon Cancer AJCC v8; Stage IV Rectal Cancer AJCC v8; Stage IVA Colon Cancer AJCC v8; Stage IVA Rectal Cancer AJCC v8; Stage IVB Colon Cancer AJCC v8; Stage IVB Rectal Cancer AJCC v8
Keywords: colon cancer; rectal cancer; colorectal cancer; microsatellite instability; circulating tumor DNA; metastasis; Immunotherapy
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Metastasis; Rectal Neoplasms; Colorectal Neoplasms; Microsatellite Instability | interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (M7824) (Experimental): Patients receive M7824 IV over 1 hour on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity (Cohorts A,B, and C) or for six doses in patients with detectable circulating tumor DNA (ctDNA) following resection of all known liver metastases (Cohort D).
  Interventions: Biological: Anti-PD-L1/TGFbetaRII Fusion Protein M7824

INTERVENTIONS:
Biological: Anti-PD-L1/TGFbetaRII Fusion Protein M7824 — Given IV
  Other Names: Anti-PDL1/TGFb Trap MSB0011359C; M7824; MSB0011359C; Bintrafusp Alfa

SUMMARY:
This phase Ib/II trial studies how well anti-PD-L1/TGFbetaRII fusion protein M7824 (M7824) works in treating patients with colorectal cancer (or with other solid tumors with microsatellite instability) that has spread to other places in the body or cannot be removed by surgery. Immunotherapy with monoclonal antibodies, such as M7824, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

-Objective response rate (ORR) in microsatellite instability-high (MSI-H) mCRC patients who have progressed on immune checkpoint blockade therapy (Cohort A).

OR

-ORR in patients with treatment-refractory, consensus molecular subtype 4 (CMS4) mCRC patients coadmnistered SBRT (Cohort B).

OR

* ORR in patients with MSI-H non CRC solid tumors who have progressed on immune checkpoint blockade therapy (Cohort C) OR
* Clearance of ctDNA in ctDNA(+) patients with resected mCRC following completion of standard-of-care therapy (Cohort D).

SECONDARY OBJECTIVES:

To estimate progression-free survival (PFS) for M7824 in patients with:

-MSI-H mCRC whose disease has progressed on prior immune checkpoint blockade therapy (Cohort A).

OR

-Treatment-refractory, CMS4 mCRC coadministered SBRT (Cohort B). While SBRT is preferred, IMRT or 3D conformal techniques may be utilized at the discretion of the treating radiation oncologist depending on the dose to surrounding normal tissues. Patient will receive a total dose of 24Gy over three days with one of the following modalities, at the discretion of the treating radiation oncologist: SBRT, IMRT and 3D conformal.

OR o MSI-H LA/UR/metastatic non-CRC solid tumors with prior progression on an immune checkpoint blockade therapy (Cohort C).

To estimate overall survival (OS) for M7824 in patients with:

o MSI-H mCRC who are refractory to prior immune checkpoint blockade therapy (Cohort A).

OR o Treatment-refractory, CMS4 mCRC coadministered SBRT (Cohort B). While SBRT is preferred, IMRT or 3D conformal techniques may be utilized at the discretion of the treating radiation oncologist depending on the dose to surrounding normal tissues. Patient will receive a total dose of 24Gy over three days with one of the following modalities, at the discretion of the treating radiation oncologist: SBRT, IMRT and 3D conformal.

OR

* MSI-H LA/UR/metastatic non-CRC solid tumors with prior progression on an immune checkpoint blockade therapy (Cohort C) OR
* ctDNA(+) resected mCRC following completion of standard-of-care therapy (Cohort D).

To estimate disease-free survival (DFS) in patients with resected mCRC following standard-of-care treatment (cohort D).

To evaluate safety and tolerability of treatment with M7824 in patients with:

o MSI-H mCRC who are refractory to prior immune checkpoint blockade therapy (Cohort A).

OR

* Treatment-refractory, CMS4 mCRC (Cohort B) OR
* MSI-H LA/UR/metastatic non-CRC solid tumors with prior progression on an immune checkpoint blockade therapy (Cohort C) OR
* ctDNA(+) resected mCRC following completion of standard-of-care therapy (Cohort D).

EXPLORATORY OBJECTIVES:

1. To evaluate intratumoral pharmacodynamic changes in immune populations using paired biopsies from patients with MSI-H solid tumors (Cohorts A and C) or CMS4 mCRC treated with M7824 and SBRT (Cohort B). While SBRT is preferred, IMRT or 3D conformal techniques may be utilized at the discretion of the treating radiation oncologist depending on the dose to surrounding normal tissues. Patient will receive a total dose of 24Gy over three days with one of the following modalities, at the discretion of the treating radiation oncologist: SBRT, IMRT and 3D conformal.
2. To characterize circulating immune cell populations and cytokine profiles in tumor and circulation following treatment with M7824.
3. To describe changes in levels of TGF-β following treatment with M7824.
4. To correlate the presence of microsatellite instability with CMS1 profile.
5. To correlate MSI-H and CMS4 to CpG island methylator phenotype (CIMP) status, KRAS and BRAF mutation status.
6. To quantify correlation with CMS4 and immune populations within tumor infiltrate.
7. To correlate anti-tumor response to M7824 with PD-L1 expression.
8. To conduct RNAseq, RNA Scope, WES targeted sequencing and tissue IO gene expression by Nanostring.
9. To evaluate novel markers in blood by liquid biopsy including, but not limited to, circulating-free DNA (cfDNA), exosomes, and circulating tumor cells (CTC).
10. To describe changes in microbiome profiling upon treatment with M7824 (with or without radiation).

OUTLINE:

For cohorts A, B, and C, patients receive M7824 intravenously (IV) over 1 hour on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

For cohort D, patients receive M7824 intravenously (IV) over 1 hour on days 1 and 15 for a total of six treatments.

After completion of study treatment, patients are followed up at 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the colon or the rectum that is metastatic or unresectable (cohorts A,B); histologically or cytologically confirmed carcinoma not originating in the colon or rectum (cohort C); or histologically or cytologically confirmed adenocarcinoma of the colon or the rectum following resection of the primary tumor and metastatic disease, following completion of standard-of-care perioperative therapy at the discretion of the treating provider (cohort D).
* Confirmation of: a) Cohort A: microsatellite instability in colorectal cancer (CRC); b) Cohort B: CMS4 CRC classification on pretreatment primary tumor; c) Cohort C: microsatellite instability in non-CRC solid tumor; d. Cohort D: microsatellite stability.
* Ability to provide written informed consent.
* Documented progression to prior therapies (Cohorts A, B, and C): a) Cohort A: Disease progression following prior immune checkpoint blockade therapy; b) Cohort B: Progression or intolerance to at least 2 prior lines of standard therapy for unresectable or metastatic CRC; c) Cohort C: Disease progression following prior immune checkpoint blockade therapy.
* Available primary tumor tissue for CMS4 biomarker assessment.
* Life expectancy >= 12 weeks as judged by the treating physician.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1(Cohorts A, B, and C). For cohort B, measureable lesions must be identified apart from the irradiated tumor lesion. Patients in cohort D must have no evidence of radiographically evident disease at the time of study entry.
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (in absence of blood transfusion).
* Lymphocyte count >= 0.5 x 10^9/L (in absence of blood transfusion).
* Platelet count >= 100 x 10^9/L (in absence of blood transfusion).
* Hemoglobin (Hgb) >= 9 g/dL (in absence of blood transfusion).
* Total bilirubin level =< 1.5 x the upper limit of normal (ULN).
* An aspartate aminotransferase (AST) level =< 2.5 x ULN, and an alanine aminotransferase (ALT) level =< 2.5 x ULN. If liver metastases are present, then it is acceptable for AST level =< 5.0 x ULN, and an ALT level =< 5.0 x ULN.
* International normalized ratio (INR) < 1.5.
* An estimated creatinine clearance > 30 mL/min according to the Cockcroft-Gault formula or be measure for creatinine clearance from 24-hour urine collection.
* Highly effective contraception for both male and female subjects if the risk of conception exists. Highly effective contraception must be used 30 days prior to first trial administration, for the duration of trial treatment, and at least for 4 months after stopping trial treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this trial, the treating physician should be informed immediately.
* Ability to tolerate receipt of radiotherapy to a metastasis not adjacent to a normal dose-limiting structure, at the discretion of the treating radiation oncologist (cohort B).
* Presence of detectable ctDNA following completion of R0 resection with or without perioperative therapy, with confirmation of somatic mutations in the resected tumor (cohort D only).
* Completion of all standard-of-care adjuvant therapy (cohort D).

Exclusion Criteria:

* Concurrent treatment with non-permitted drugs and other interventions.
* Anticancer treatment within 14 days before the start of trial treatment (e.g., cytoreductive therapy, radiotherapy [with the exception of palliative radiotherapy delivered in a normal organ-sparing technique], immune therapy, or cytokine therapy).
* Major surgery as determined by the investigator within 28 days before the start of trial treatment (prior diagnostic biopsy is permitted).
* Systemic therapy with immunosuppressive agents within 7 days before the start of treatment; or use of any investigational drug within 28 days before the start of trial treatment.
* Cohort A and C only: Intolerance or serious adverse immune related adverse events (irAEs) that were symptomatic or required or continues to require ongoing immunosuppression to previous immune checkpoint therapy.
* Cohort B and D: prior exposure to any immune checkpoint blockade agent or any other immunomodulatory agent used for antineoplastic therapy for mCRC.
* Previous malignant disease (other than the target malignancy to be investigated in this trial) within 3 years prior to study treatment initiation. Subjects with a history of cervical carcinoma in situ, superficial or non-invasive bladder cancer, or basal cell or squamous cell carcinoma in situ, previously treated with curative intent are NOT excluded. Subjects with other localized malignancies treated with curative intent need to be discussed with the principal investigator.
* Subjects with active central nervous system (CNS) metastases are excluded. Subjects with a history of treated CNS metastases (by surgery or radiation therapy) are not eligible unless they have fully recovered from treatment, demonstrated no progression for at least 2 months, and do not require continued steroid therapy.
* Receipt of any organ transplantation, including allogeneic stem-cell transplantation, but with the exception of transplants that do not require immunosuppression (e.g., corneal transplant, hair transplant).
* Significant acute or chronic infections including, among others: a) Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome; b) Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (HBV surface antigen positive and HBV core antibody positive with reflex to positive HBV DNA or HBV core antibody positive alone with reflex to positive HBV DNA or positive HCV antibody with reflex to positive HCV ribonucleic acid [RNA]); c) Subjects with active tuberculosis (history of exposure or history of positive tuberculosis test plus presence of clinical symptoms, physical or radiographic findings).
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent: a) Subjects with type I diabetes, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible; b) Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses =< 10 mg of prednisone or equivalent per day; c) Administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable.
* Known severe hypersensitivity reactions to monoclonal antibodies (grade >= 3 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE] v4.03), any history of anaphylaxis, or recent (within 5 months) history of uncontrolled asthma.
* Persisting toxicity (except alopecia and vitiligo) related to prior oncologic therapy grade > 1 NCI-CTCAE v4.03, however, sensory neuropathy grade =< 2 is acceptable.
* Clinically significant cardiovascular/ cerebrovascular disease as follows: cerebral vascular accident / stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification class > II), or serious cardiac arrhythmia.
* Clinically relevant diseases (for example, inflammatory bowel disease) and / or uncontrolled medical conditions, which, in the opinion of the Investigator, might impair the subject's tolerance or ability to participate in the trial.
* Vaccine administration within 4 weeks of M7824 administration. Vaccination with live vaccines while on trial is prohibited. Administration of inactivated vaccines is allowed (for example, inactivated influenza vaccines).
* Cohort D: peritoneal carcinomatosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Van K Morris, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Morris JS, Luthra R, Liu Y, Duose DY, Lee W, Reddy NG, Windham J, Chen H, Tong Z, Zhang B, Wei W, Ganiraju M, Broom BM, Alvarez HA, Mejia A, Veeranki O, Routbort MJ, Morris VK, Overman MJ, Menter D, Katkhuda R, Wistuba II, Davis JS, Kopetz S, Maru DM. Development and Validation of a Gene Signature Classifier for Consensus Molecular Subtyping of Colorectal Carcinoma in a CLIA-Certified Setting. Clin Cancer Res. 2021 Jan 1;27(1):120-130. doi: 10.1158/1078-0432.CCR-20-2403. Epub 2020 Oct 27. PMID 33109741
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective, single-arm pilot study of BA as monotherapy conducted under Institutional Review Board approval at The University of Texas MD Anderson Cancer Center (Houston, TX).
Groups:
- IV Bintrafusp Alfa Every 14 Days at a Fixed Dose of 1200 mg: 6 planned doses until one of the following events (whichever came first): therapeutic failure requiring urgent additional antineoplastic therapy, unacceptable toxicity, onset of pregnancy, or withdrawal of informed consent. Followed by evaluation for treatment response with repeat ctDNA analysis.
Period: Overall Study
Arm/Group | IV Bintrafusp Alfa Every 14 Days at a Fixed Dose of 1200 mg
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IV Bintrafusp Alfa Every 14 Days at a Fixed Dose of 1200 mg
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 55.9 [42.5 to 68.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Circulating DNA Clearance
Description: Defined as the percentage of somatic mutations, ctDNA that is eliminated in blood as well as no appearance of any new somatic mutations following six doses of BA in the study participants.
Time Frame: Baseline up to 12 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of DNA cleared
Arm/Group | IV Bintrafusp Alfa Every 14 Days at a Fixed Dose of 1200 mg
Number analyzed (Participants) | 4
percentage of DNA cleared | 0 [0 to 60]

2. Secondary Outcome: Overall Survival (OS)
Description: Number of participants alive from baseline through 2 years
Time Frame: Baseline up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | IV Bintrafusp Alfa Every 14 Days at a Fixed Dose of 1200 mg
Number analyzed (Participants) | 4
Participants | 4

3. Secondary Outcome: Grade 3 or Higher A/E Per CTCAE v4.03
Description: The occurrence of grade 3 or higher adverse events according to CTCAE version 4.03
Time Frame: Start of study treatment up to 28 days after end of treatment
Measure: Number; unit: number of events
Arm/Group | IV Bintrafusp Alfa Every 14 Days at a Fixed Dose of 1200 mg
Number analyzed (Participants) | 4
number of events | 0

4. Secondary Outcome: Disease-Free Survival (DFS)
Description: The time from the date of first administration of BA until the date of documented recurrence or development of distant metastasis by RECIST.
Time Frame: Baseline up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | IV Bintrafusp Alfa Every 14 Days at a Fixed Dose of 1200 mg
Number analyzed (Participants) | 4
Months | 3 [0.9 to 27]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | IV Bintrafusp Alfa Every 14 Days at a Fixed Dose of 1200 mg
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Bintrafusp Alfa Every 14 Days at a Fixed Dose of 1200 mg (N=4)
Rash (Skin and subcutaneous tissue disorders) | 3
Squamous Cell Ca of the Skin (Skin and subcutaneous tissue disorders) | 1
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Condyloma (Skin and subcutaneous tissue disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine Kinase Increased (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Flu-Like Symptoms (General disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT03436563/Prot_SAP_000.pdf